CLINICAL TRIAL: NCT04069104
Title: Whack-a-Mole: Testing an Intervention to Increase Melanoma Identification
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Nicholas Carcioppolo, Associate Professor, University of Miami
Other Study IDs: 20190153
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Diagnoses Disease
Keywords: Melanoma identification

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- ABCD training with standard feedback: Asymmetry, Border, Color, Diameter (ABCD) training message intervention with standard dermatological feedback
  Interventions: Behavioral: ABCD Information; Behavioral: Standard (clinical) feedback
- ABCD training with motivational feedback: ABCD training message intervention with dermatological feedback and a motivational message
  Interventions: Behavioral: ABCD Information; Behavioral: Motivational feedback
- ABCD training with no feedback: ABCD message intervention with no feedback
  Interventions: Behavioral: ABCD Information
- UDS method training with standard feedback: Ugly Duckling Sign (UDS) method message intervention with dermatological feedback.
  Interventions: Behavioral: UDS information; Behavioral: Standard (clinical) feedback
- UDS method training with motivational feedback: UDS message intervention with dermatological feedback and a motivational message.
  Interventions: Behavioral: UDS information; Behavioral: Motivational feedback
- UDS training with no feedback: UDS message intervention with no feedback.
  Interventions: Behavioral: UDS information
- ABCD-F training with standard feedback: ABCD-F intervention with dermatological feedback.
  Interventions: Behavioral: ABCD Information; Behavioral: UDS information; Behavioral: Standard (clinical) feedback
- ABCD-F training with motivational feedback: ABCD-F intervention with dermatological feedback and a motivational message.
  Interventions: Behavioral: ABCD Information; Behavioral: UDS information; Behavioral: Motivational feedback
- ABCD-F training with no feedback: ABCD-F intervention with no feedback.
  Interventions: Behavioral: ABCD Information; Behavioral: UDS information
- No message intervention with standard feedback: No message intervention, but with dermatological feedback.
  Interventions: Behavioral: Standard (clinical) feedback
- No message intervention with motivational feedback: No message intervention, but with dermatological feedback and a motivational message.
  Interventions: Behavioral: Motivational feedback
- No message intervention with no feedback: No message intervention and no feedback. True control.

INTERVENTIONS:
Behavioral: ABCD Information — The intervention condition includes exposure to a message emphasizing the ABCD strategy to identify malignant melanoma.
  Groups: ABCD training with motivational feedback; ABCD training with no feedback; ABCD training with standard feedback; ABCD-F training with motivational feedback; ABCD-F training with no feedback; ABCD-F training with standard feedback
Behavioral: UDS information — The intervention condition includes exposure to a message emphasizing the UDS strategy to identify malignant melanoma.
  Groups: ABCD-F training with motivational feedback; ABCD-F training with no feedback; ABCD-F training with standard feedback; UDS method training with motivational feedback; UDS method training with standard feedback; UDS training with no feedback
Behavioral: Standard (clinical) feedback — Feedback on mole identification task provided by a dermatologist.
  Groups: ABCD training with standard feedback; ABCD-F training with standard feedback; No message intervention with standard feedback; UDS method training with standard feedback
Behavioral: Motivational feedback — Feedback on mole identification task provided by a dermatologist plus exposure to a motivational fear appeal message designed to increase skin self exam intentions.
  Groups: ABCD training with motivational feedback; ABCD-F training with motivational feedback; No message intervention with motivational feedback; UDS method training with motivational feedback

SUMMARY:
The purpose of this study is to evaluate an interactive game designed to increase people's ability to identify cancerous moles.

ELIGIBILITY:
Inclusion Criteria:

* Resident of U.S.
* At least 18 years old
* Capable of reading English
* Member of panel assembled by survey provider

Exclusion Criteria:

* Individuals under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults living in U.S. who are members of the online panel.
Sampling Method: Probability Sample
Enrollment: 1849 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Mole identification accuracy | Day 2
  Mole identification accuracy will be reported as the amount of mole correctly identified as either melanoma or typical nevi

SECONDARY OUTCOMES:
Skin Self Exam Intentions | Day 2
  Self-report measure of intentions to perform a skin self exam. Quantified using a single item indicator with scores ranging from 1-7 with higher scores indicating greater intentions to perform a skin self exam to detect potential melanomas.
Intentions to see a Dermatologist | Day 2
  Self-report measure of intentions to schedule an appointment with a dermatologist to receive a skin cancer exam. Quantified using a single item indicator with scores ranging from 1-7 with higher scores indicating greater intentions to schedule an appointment with a dermatologist.
Skin Self Exam Attitudes | Day 2
  Self-report measure of attitudes towards skin cancer exams. Quantified using the mean of the self report scale with scores ranging from 1-7 with higher scores indicating more positive attitudes towards skin self exams.
Skin Self Exam Beliefs | Day 2
  Self-report measure of beliefs towards skin cancer exams. Quantified using the mean of the self report scales for perceived susceptibility, perceived severity, perceived self-efficacy, and perceived response efficacy with scores ranging from 1-7 with higher scores indicating more strongly held beliefs about skin self exams.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Carcioppolo, PhD, Principal Investigator — Study Co-Principal Investigator; Soyoon Kim, PhD, Principal Investigator — Study Co-Principal Investigator
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No